CLINICAL TRIAL: NCT02124304
Title: EMG Activation of Cervical Musculature During Therapeutic Exercise With Thera-Band(R) Resistance Versus Manual Resistance
Brief Title: Cervical Activation During Elastic and Manual Resistance
Acronym: CervEMG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sport and Spine Rehab Clinical Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SSR04
Record Dates: First submitted 2014-04-22; First posted 2014-04-28 (Estimated); Results first posted 2016-02-09 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-01

CONDITIONS: Cervical Pain
Keywords: Sternocleidomastoid; Neck pain; EMG; Perceived Exertion; Thera-Band; Cervical Paraspinals
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cervical Pain (Experimental): Thera-Band elastic and manual resistance neck exercises for neck strengthening
  Interventions: Device: Neck exercises using both manual and Thera-Band elasatic resistance
- Healthy (Experimental): Thera-Band elastic and manual resistance neck exercises for neck strengthening
  Interventions: Device: Neck exercises using both manual and Thera-Band elasatic resistance

INTERVENTIONS:
Device: Neck exercises using both manual and Thera-Band elasatic resistance — Exercises will include cervical flexion and extension, and cervical right and left side-bending, and rotation. All 6 exercises will be done with both manual and elastic (Thera-Band) resistance.Manual Resistance is applied by the subject placing their own hand on their head and pushing in to it. Thera-Band bands will be used to provide elastic resistance
  Other Names: Thera-Band

SUMMARY:
Cervical pain is a condition that affects 14.6% of all adults annually. Of this annual prevalence, 37.3% experience persistent neck pain with periodic recurring episodes. The purpose of this study is to compare muscle activation patterns of the cervical musculature during exercises with elastic versus manual resistance in a neck pain and asymptomatic populations. Methods: A convenience sample of 15 healthy, physically active participants and 15 current patients diagnosed with non-radicular cervical pain will be recruited. Exclusionary criteria will include: current cervical or upper extremity injury (healthy group), history of neck surgery, corticosteroid treatment within the last two weeks, and radicular signs or symptoms. Surface electromyography will be used to quantify the activity level of the bilateral SCM, AS, Cervical Paraspinal (CP), and the Upper Trapezius (UT) muscles while performing a series of 6 exercises with elastic resistance using Thera-Band® Resistance Bands and manual resistance. The area will be prepped and surface electrodes placed on the corresponding muscles. The movement will be standardized by using the peak activation (PA) of each muscle during full flexion-extension movement to create a percentage of peak activation (%PA). The testing battery will consist of 6 exercises with elastic resistance and manual resistance, totaling 12 different trials. Each trial will involve 5 repetitions, each held for 5 seconds. The exercises will include cervical: extension, flexion, left rotation, right rotation, left side bending, and right side bending. The men will use the green and women will use the red Thera-Band® Resistance Band. The order of exercises will be randomized in to two parts to minimize the effect of fatigue. First, cervical flexion and extension with manual and elastic resistance will be randomized. Secondly, the remaining 8 exercises will be randomized. Following each exercise, the patient will rate their perceived level of exertion on the Thera-band® Resistance Intensity Scale for Exercise (RISE).

ELIGIBILITY:
Inclusion Criteria:

* healthy physically active subjects (healthy group)
* patients diagnosed with non-radicular cervical neck pain (neck pain group)
* 18-65

Exclusion Criteria:

* current cervical or upper extremity injury (healthy group)
* history of neck surgery
* corticosteroid treatment within the last two weeks
* radicular signs or symptoms

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-04; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barton Bishop, DPT, Principal Investigator — Sport & Spine Rehab Clinical Research Foundation
Locations (1):
- Sport & Spine Rehab, Rockville, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Cervical Neck Pain; Healthy: Thera-Band elastic and manual resistance neck exercises for neck strengthening
  Neck exercises using both manual and Thera-Band elasatic resistance: Exercises will include cervical flexion and extension, and cervical right and left side-bending, and rotation. All 6 exercises will be done with both manual and elastic (Thera-Band) resistance.Manual Resistance is applied by the subject placing their own hand on their head and pushing in to it. Thera-Band bands will be used to provide elastic resistance
Period: Overall Study
Arm/Group | Cervical Neck Pain | Healthy
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cervical Neck Pain | Healthy | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Full Range); unit: years] | 31.8 [24 to 47] | 28.1 [21 to 36] | 29.95 [21 to 47]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 6 | 9 | 15

OUTCOME MEASURES:

1. Primary Outcome: Percent of Peak Activation (%PA)
Description: 8 muscles during 12 exercises were analyzed in 30 subjects, totaling 2880 data points. At the beginning of the study, peak activation (PA) was assessed for each muscle during full flexion-extension, used as a reference exercise. For each subject, the EMG signals of the muscles during the 12 exercises were smoothed, rectified and analyzed using a root-mean-square algorithm and the greatest activation of each muscle was used. After the PA for each muscle was determined, it was compared to the PA of the reference exercise for the respective muscle group, and expressed as a percent of the peak activation (%PA). In some cases the %PA is greater than 100%. This is possible as the PA was assessed during a full flexion-extension movement. During an exercise some muscles generated greater PA and therefore when the calculations were performed the %PA was greater than 100%. Due to the extensive amount of data, we have provided the Left Cervical Paraspinals %PA results for each exercise.
Time Frame: One 1 hour session
Measure: Mean (Full Range); unit: Percentage of Peak Activation (%PA)
Arm/Group | Cervical Pain | Healthy
Number analyzed (Participants) | 15 | 15
Percentage of Peak Activation (%PA)
  Flexion Manual | 51.72 [20.89 to 92.37] | 61.20 [40.79 to 107.94]
  Extension Manual | 88.1 [32.62 to 217.92] | 80.80 [43.7 to 156.61]
  Flexion Elastic | 65.68 [20.61 to 152.75] | 86.81 [33.54 to 129.10]
  Extension Elastic | 60.60 [28.98 to 115.07] | 71.9 [39.59 to 137.28]
  Right Rotation Manual | 61.02 [11.93 to 152.75] | 68.99 [22.63 to 163.92]
  Left Rotation Manual | 108.44 [33.33 to 220.39] | 180.20 [66.67 to 694.44]
  Right Rotation Elastic | 61.45 [21.55 to 126.27] | 70.70 [27.22 to 146.60]
  Left Rotation Elastic | 81.53 [30.86 to 150.13] | 103.66 [6.94 to 264.08]
  Right SideBending Manual | 62.33 [23.63 to 144.91] | 66.48 [5.33 to 115.91]
  Left SideBending Manual | 100.10 [35.07 to 284.21] | 115.60 [32.89 to 191.96]
  Right SideBending Elastic | 57.66 [19.02 to 142.30] | 65.69 [32.21 to 131.06]
  Left SideBending Elastic | 55.44 [23.2 to 155.35] | 84.95 [55.53 to 119.63]

2. Secondary Outcome: Perceived Exertion
Description: Thera-Band(R) RISE (Resistance Intensity Scale for Exercise) Scale to measure amount of perceived exertion during resistance band exercises. Participants were asked to rate the intensity of an exercise on a scale from 0 to 10, 0 being no resistance and 10 being the maximum resistance.
Time Frame: 12 exercises during one 1 hour session
Measure: Mean (Full Range); unit: units on a scale, ranging from 0 to 10
Arm/Group | Cervical Pain | Healthy
Number analyzed (Participants) | 15 | 15
units on a scale, ranging from 0 to 10
  Flexion Manual | 4.9 [0 to 10] | 4.1 [1 to 7]
  Extension Manual | 3.5 [0 to 7] | 3.5 [1 to 7]
  Flexion Elastic | 4.6 [1 to 8] | 4.5 [1 to 8]
  Extension Elastic | 4.1 [1 to 9] | 3.3 [0 to 6]
  Right Rotation Manual | 4.5 [0 to 10] | 3.5 [0 to 7]
  Left Rotation Manual | 4.5 [0 to 10] | 3.3 [0 to 6]
  Right Rotation Elastic | 3.4 [0 to 6] | 3.1 [0 to 6]
  Left Rotation Elastic | 4 [1 to 6] | 3.1 [0 to 6]
  Right SideBending Manual | 4.6 [0 to 9] | 3.9 [1 to 9]
  Left SideBending Manual | 3.9 [0 to 8] | 3.5 [1 to 6]
  Right SideBending Elastic | 4.1 [0 to 10] | 3.5 [1 to 6]
  Left SideBending Elastic | 4.1 [0 to 8] | 3.2 [1 to 6]

ADVERSE EVENTS:
Arm/Group | Cervical Neck Pain | Healthy
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No